CLINICAL TRIAL: NCT03300531
Title: Autologous Pure Platelet-rich Plasma in the Treatment of Tendon Disease：A Randomized Controlled Trial
Brief Title: Impact of Autologous Pure Platelet-rich Plasma in the Treatment of Tendon Disease
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Collaborators: Zhejiang Xingyue Biotechnology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2017.N0.003
Record Dates: First submitted 2017-09-28; First posted 2017-10-03 (Actual); Last update posted 2017-10-09 (Actual); Status verified 2017-09

CONDITIONS: Rotator Cuff Tear; Lateral Epicondylitis; Achilles Tendinitis
Keywords: Pure Platelet-rich Plasma; Randomized Controlled Trial
MeSH Terms: conditions — Rotator Cuff Injuries; Tennis Elbow | interventions — Injections

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- P-PRP (Experimental): Blood will be drawn and pure platelet-rich plasma will be injected into the tendon.
  Interventions: Biological: Ultrasound-guided pure platelet-rich-plasma (P-PRP) injection
- PRP (Experimental): Blood will be drawn and platelet-rich plasma will be injected into the tendon.
  Interventions: Biological: Ultrasound-guided platelet-rich-plasma (PRP) injection
- Compound betamethasone (Active Comparator): 1ml dexamethasone mixed with 0.5-2ml of saline to achieve the same injection volume (which contains betamethasone dipropionate 5mg and betamethasone sodium phosphate 2mg) )
  Interventions: Drug: Ultrasound-guided Compound betamethasone injection

INTERVENTIONS:
Biological: Ultrasound-guided pure platelet-rich-plasma (P-PRP) injection — Blood will be drawn, and tendon will be penetrated with dry needle under ultrasound guidance. Pure platelet-rich plasma will be injected into the tendon.Once a week for three times.
  Arms: P-PRP
Biological: Ultrasound-guided platelet-rich-plasma (PRP) injection — Blood will be drawn, and tendon will be penetrated with dry needle under ultrasound guidance. Platelet-rich plasma will be injected into the tendon.Once a week for three times.
  Arms: PRP
Drug: Ultrasound-guided Compound betamethasone injection — Tendon will be penetrated with dry needle under ultrasound guidance. Compound betamethasone will be injected into the tendon.Once a week for three times.
  Arms: Compound betamethasone

SUMMARY:
This is a randomized parallel controlled double-blind phase 2 clinical study.All subjects are recruited from the patients of rotator cuff tear, lateral epicondylitis or chronic achilles tendonitis. Patients will be randomly divided into three groups. Autologous pure platlet-rich plasma (P-PRP) and platlet-rich plasma (PRP) are purified from the peripheral blood .Patients of case groups will receive P-PRP or PRP injection once a week for three times while the control group received the same dose compound betamethasone injection. Follow up visit will occur at 1 month,3 months, 6 months,12 months after the last injection. Clinical quantitative assessment will measure by the visual analogue scale(VAS). The secondary outcomes are the constant-murley score(CMS) and the rating scale of the American shoulder and elbow surgeons(ASES) and the disability of arm shoulder and hand(DASH). The objective evaluation methods is that the examination of MRI or ultrasound were accomplished before the first injection and at 6 and 12 months afterwards.

DETAILED DESCRIPTION:
All injection will be done under ultrasound guidance.

ELIGIBILITY:
Inclusion Criteria:

1. clinically diagnosed as rotator cuff tear, lateral epicondylitis or chronic achilles tendonitis;
2. symptom duration is over 3 months, non-steroidal drug treatment , rehabilitation treatment and other conservative treatment is invalid;
3. patient that can understand the clinical trials and signed the informed consent.

Exclusion Criteria:

1. patient that underwent other injection treatment within 6 weeks
2. some associated diseases (such as arthritis, synovitis, entrapment of related nerve, radiculopathy to the target lesion, generalized pain syndrome, rheumatoid arthritis, pregnancy, impaired sensibility, paralysis, history of allergic or hypersensitive reaction to bovine-derived proteins or fibrin glue)
3. patient that enrolled other clinical trials within 3 months
4. history of drug/alcohol addiction, habitual smoker

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 540 (Estimated)
Dates: Start 2017-12-01 (Estimated); Primary Completion 2020-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in Visual Analog Scale(VAS) at 3, 6 and 12 weeks | Baseline, 3 weeks, 6 weeks, 12 weeks after intervention
  Pain on activity will be evaluated by VAS

SECONDARY OUTCOMES:
Constant-Murley Score(CMS) | Baseline, 3 weeks, 6 weeks, 12 weeks after intervention
  Functional score of the shoulder
American Shoulder and Elbow Surgeons (ASES) Shoulder Score | Baseline, 3 weeks, 6 weeks, 12 weeks after intervention
  Functional score of the shoulder
The Disabilities of the Arm, Shoulder and Hand(DASH) Score | Baseline, 3 weeks, 6 weeks, 12 weeks after intervention
  Functional score of the shoulder
Victorian Institute of Sport Assessment-Achilles questionnaire (VISA-A) | Baseline, 3 weeks, 6 weeks, 12 weeks after intervention
  Functional score of the achilles tendon
Adverse events | From baseline through study completion, an average of 3 year
  Adverse events to evaluate the safety

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Karjalainen TV, Silagy M, O'Bryan E, Johnston RV, Cyril S, Buchbinder R. Autologous blood and platelet-rich plasma injection therapy for lateral elbow pain. Cochrane Database Syst Rev. 2021 Sep 30;9(9):CD010951. doi: 10.1002/14651858.CD010951.pub2. PMID 34590307